CLINICAL TRIAL: NCT03800290
Title: Targeting the Beta-2-adrenergic Pathway to Improve Skeletal Muscle Glucose Uptake in Healthy Humans
Brief Title: Human Beta-2 Adrenergic Stimulation and Muscle Glucose Uptake
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NL67646.068.18
Record Dates: First submitted 2018-12-06; First posted 2019-01-11 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: Beta-2 adrenergic agonist; Glucose homeostasis; Skeletal muscle; Human

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, cross-over, single-center study
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clenbuterol hydrochloride (Experimental): Subjects will ingest clenbuterol hydrochloride capsules (20 microgram/each) twice daily (40 microgram/day) for a maximum of 14 days.
  Subjects that received the clenbuterol hydrochloride capsules (at random) in the first study period will receive the placebo capsules during the second study period.
  Interventions: Drug: Clenbuterol Hydrochloride
- Placebos (Placebo Comparator): Subjects will ingest placebo capsules matching the clenbuterol hydrochloride capsules one time per day for a maximum of 14 days.
  Subjects that received the placebo capsules (at random) in the first study period will receive the clenbuterol hydrochloride capsules during the second study period.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Clenbuterol Hydrochloride — Daily ingestion of clenbuterol hydrochloride capsules (40 microgram/day) for a total period of 14 days with a wash-out period of 4 weeks.
  Arms: Clenbuterol hydrochloride
Drug: Placebos — Daily ingestion of placebo capsules for a total period of 14 days with a wash-out period of 4 weeks.
  Arms: Placebos

SUMMARY:
The purpose of this study is to investigate the effect of two weeks clenbuterol/placebo supplementation on skeletal muscle glucose disposal in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian;
2. Male sex;
3. Age: 18-30
4. BMI: 18-25 kg/m2;
5. Normal physical activity levels;

Exclusion Criteria:

1. Not meeting all inclusion criteria
2. Cardiovascular diseases (determined by means of questionnaires, heart rate/blood pressure measurements)
3. Respiratory diseases (including asthma, bronchitis and COPD);
4. Unstable body weight (weight gain or loss > 5 kg in the last three months);
5. Intention to lose or gain body weight (e.g. with caloric restriction or physical activity)
6. Excessive alcohol and/or drug abuse;
7. Hypokalaemia;
8. Hb < 8.4 mmol/L;
9. Epilepsy;
10. Smoking;
11. Renal and/or liver insufficiency;
12. Participation in another biomedical study within 1 month before the first study visit, possibly interfering with the study results;
13. Medication use known to hamper subject's safety during the study procedures;
14. Subjects who do not want to be informed about unexpected medical findings;
15. Subjects who do not want that their treating physician to be informed;
16. Inability to participate and/or complete the required measurements;
17. Participation in organised or structured physical exercise;
18. Any condition, disease or abnormal laboratory test result that, in the opinion of the Investigator, would interfere with the study outcome, affect trial participation or put the subject at undue risk;
19. Hyperthyroidism

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Insulin-stimulated peripheral glucose disposal (Rd) | 2 weeks
  Comparison between prolonged (2 weeks) clenbuterol hydrochloride or placebo supplementation on insulin-stimulated peripheral glucose disposal (Rd) during the high-insulin infusion step during the two-step hyperinsulinemic-euglycemic clamp.

SECONDARY OUTCOMES:
Skeletal muscle GLUT4 translocation | acute (4 hours) and long-term (2 weeks)
  Comparison between acute (4h) and prolonged (2 weeks) clenbuterol hydrochloride or placebo supplementation on skeletal muscle GLUT4 translocation as assessed by means of wide-field microscopy in skeletal muscle biopsies

OTHER OUTCOMES:
Body weight/composition | 2 weeks
  Comparison between prolonged (2 weeks) clenbuterol hydrochloride or placebo supplementation on body weight and composition as assessed by means of a Bodpod measurement.
Plasma substrates | Acute (4 hours) and long-term (1 and 2 weeks)
  Comparison between acute (4h) and prolonged (1 and 2 weeks) clenbuterol hydrochloride or placebo supplementation on plasma substrate concentrations, including insulin, glucose, free fatty acids and TAGs.
Heart rate | Acute (4 hours) and long-term (1 and 2 weeks)
  Comparison between acute (4h) and prolonged (1 and 2 weeks) clenbuterol hydrochloride or placebo supplementation on heart rate as measured by means of an automated cuff.
Blood pressure | Acute (4 hours) and long-term (1 and 2 weeks)
  Comparison between acute (4h) and prolonged (1 and 2 weeks) clenbuterol hydrochloride or placebo supplementation on blood pressure (systolic and diastolic) as measured by means of an automated cuff.
Insulin-mediated suppression of hepatic glucose production | 2 weeks
  Comparison between prolonged (2 weeks) clenbuterol hydrochloride or placebo supplementation on hepatic glucose production as assessed during the two-step hyperinsulinemic-euglycemic clamp.
Energy expenditure and substrate oxidation | Acute (4 hours) and long-term (2 weeks)
  Comparison between acute (4h) and prolonged (2 weeks) clenbuterol hydrochloride or placebo supplementation on energy expenditure and substrate oxidation as assessed by means of indirect calorimetry.
Sleeping energy expenditure and substrate oxidation | 2-weeks
  Comparison between prolonged (2 weeks) clenbuterol hydrochloride or placebo supplementation on sleeping energy expenditure and substrate oxidation as assessed by means of a metabolic chamber (indirect calorimetry).
Skeletal muscle glycogen | 2 weeks
  Comparison between prolonged (2 weeks) clenbuterol hydrochloride or placebo supplementation on skeletal muscle glycogen as assessed in muscle biopsies.
Skeletal muscle lipid content using wide-field microscopie | 2 weeks
  Comparison between prolonged (2 weeks) clenbuterol hydrochloride or placebo supplementation on skeletal muscle lipid content as assessed in muscle biopsies by wide-field microscopie.
Skeletal muscle gene expression | Acute (4 hours) and long-term (1 and 2 weeks)
  Comparison between acute (4h) and prolonged (2 weeks) clenbuterol hydrochloride or placebo supplementation on skeletal muscle gene expression of specific pathways as determined in muscle biopsies by means of RT-qPCR
Skeletal muscle protein expression using western blotting | Acute (4 hours) and long-term (1 and 2 weeks)
  Comparison between acute (4h) and prolonged (2 weeks) clenbuterol hydrochloride or placebo supplementation on skeletal muscle protein expression of specific pathways as determined in muscle biopsies as determined by means of Western Blotting

CONTACTS AND LOCATIONS:
Overall Officials: Joris Hoeks, PhD, Principal Investigator — principle investigator
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] van Beek SMM, Bruls YMH, Vanweert F, Fealy CE, Connell NJ, Schaart G, Moonen-Kornips E, Jorgensen JA, Vaz FM, Smeets ETHC, Joris PJ, Gemmink A, Houtkooper RH, Hesselink MKC, Bengtsson T, Havekes B, Schrauwen P, Hoeks J. Effect of beta2-agonist treatment on insulin-stimulated peripheral glucose disposal in healthy men in a randomised placebo-controlled trial. Nat Commun. 2023 Jan 12;14(1):173. doi: 10.1038/s41467-023-35798-5. PMID 36635304